CLINICAL TRIAL: NCT00100737
Title: A Phase 2 Randomized, Open-Label, Controlled Trial of the Addition of 8 Weeks SC Administration of Aldesleukin (Rh-Interleukin-2 [IL-2]) to 4 Weeks of IV Administration of Rituximab in the Treatment of Rituximab Naïve Subjects With Follicular Non-Hodgkin's Lymphoma, Refractory or Relapsed After Previous Chemotherapy
Brief Title: Comparing Interleukin-2 (IL-2) Combined With Rituximab (Rituxan) to Rituximab Alone in Subjects With Non-Hodgkin's Lymphoma (NHL)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Chiron Corporation (Industry)
Allocation: Randomized | Masking: None | Purpose: Treatment
Other Study IDs: IL2NHL006
Record Dates: First submitted 2005-01-06; First posted 2005-01-07 (Estimated); Last update posted 2006-02-06 (Estimated); Status verified 2006-02

CONDITIONS: Non-Hodgkin Lymphoma
Keywords: non-hodgkins lymphoma; interleukin-2; rituximab; CD20+ follicular B-cell non-hodgkins lymphoma (grade I, II,III)
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Lymphoma, Follicular | interventions — Interleukin-2; Rituximab

INTERVENTIONS:
Drug: interleukin-2
Drug: rituximab

SUMMARY:
The purpose of this study is to determine whether interleukin-2 given 3 times weekly for 8 weeks in combination with rituximab is effective and safe when compared to rituximab given alone in the treatment of follicular NHL subjects that have never received rituximab as a treatment and are refractory or relapsed after previous chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* CD20+ follicular B-cell non-hodgkin's lymphoma with at least 1 site of measurable disease.
* Previous treatment with 1 to 4 prior chemotherapy regimens
* ECOG performance status of greater than or equal to 2
* Life expectancy of greater than 18 weeks
* Meet safety lab requirements and organ function tests

Exclusion Criteria:

* Prior treatment with rituximab or IL-2
* Prior radioimmunotherapy including Zevalin or Bexxar
* 5 or more prior chemotherapy regimens
* Clinically significant cardiac disease, lung dysfunction, autoimmune disease, thyroid disease, active infection, unstable psychiatric condition, or HIV infection.
* History of allogenic bone marrow transplant
* Female subjects that are pregnant or breast feeding
* Immunosuppressive therapy including corticosteroids or investigational agents within 4 weeks prior to the planned start of study treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300

CONTACTS AND LOCATIONS:
Locations (1):
- Roswell Park Cancer Institute, Buffalo, New York, United States